CLINICAL TRIAL: NCT04314102
Title: The Effect of Kinesiophobia on Spatio-temporal and Functionality in Individuals Who Have Undergone Total Knee Replacement Surgery
Brief Title: The Effect of Kinesiophobia on Spatio-temporal and Functionality in Total Knee Replacement Surgery
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Furkan BİLEK, Principal Investigator, Firat University
Other Study IDs: FiratUni
Record Dates: First submitted 2020-03-13; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Kinesiophobia; Knee Osteoarthritis; Quality of Life
Keywords: knee arthroplasty; kinesiophobia; spatio-temporal; knee osteoarthritis; functionality
MeSH Terms: conditions — Kinesiophobia; Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Individuals will be evaluated before knee arthroplasty surgery. They will come for control in the 1st and 3rd months after surgery.
  No intervention will be made.
  Interventions: Other: No intervention will be made.

INTERVENTIONS:
Other: No intervention will be made. — No intervention will be made. Only checks will be made

SUMMARY:
It is stated that after arthroplasty surgery, besides the physiological factors, the factors related to the individuals may affect the recovery. Among these factors, one of the most defined in the literature is kinesiophobia. Although kinesiophobia is defined as the terms of "fear of movement" and "fear related to pain"; There are also definitions for situations in which fear of movement is most extreme or pain-related fear avoidance beliefs. Kinesiophobia, which usually occurs in the preoperative period and supports the development of chronic pain, may also affect the early recovery findings. It is very important to determine the presence and severity of kinesiophobia as it is associated with functional results after surgery.

Individuals' perceptions about themselves, expectations of recovery, and personal beliefs before surgery are thought to affect recovery in the early period. In the studies conducted, it was stated that individuals with high perception about himself and the surgical process recover faster and return to activities. However, it is emphasized that studies should be conducted on the effect of individuals' personal factors such as self-efficacy, self-perception and their perspective on health on the healing process.

DETAILED DESCRIPTION:
Osteoarthritis, which is encountered more and more with the aging population; It can occur depending on various factors such as gender, age, genetic factors, type of nutrition and joint structure. According to the studies, osteortritis ranks eleventh in the world among the factors that cause disability in individuals. Self-care activities of osteortritis individuals, especially in walking and mobility restrictions, also limit the participation of producers and leisure activities. Pain is among the most important findings that cause limitation in participation for osteoarthritis, which is frequently seen in individuals over the age of 40. In individuals with osteoarthritis, methods such as the use of non-steroidal anti-inflammatory drugs and physical rehabilitation in coping with pain are frequently used in cases where these methods are insufficient.

Total knee arthroplasty (TDA) is a surgical approach that is frequently applied to reduce pain due to severe joint damage to the knee, improve functionality and quality of life. In our country, approximately 20 thousand knee arthroplasty surgeries are performed every year and individuals who have undergone this surgery are frequently among individuals over 60 years old. This surgery is usually performed in cases of pain, deformity or severe dysfunction resulting from arthritis (osteoarthritis, rheumatoid arthritis, other). Osteoarthritis is seen as one of the main causes of this practice.

Factors such as decreased pain, increased quality of life, increased functionality and decreased level of dependence on others are among the expectations for recovery from patients after surgery. Studies show that individuals can return to daily activities for the first six weeks after surgery, and pain-related symptoms decrease in the first four weeks and therefore functional recovery is accelerated. It is stated that full recovery includes a one-year period. However, among the reasons that negatively affect post-surgical healing, various conditions ranging from systemic problems to mortality, complications due to the healing of wounds, circulatory problems, motor losses due to peroneal nerve damage, impaired biomechanics of the knee joint, development of infection, relaxation of arthroplasty, dislocations and post-surgical idiopathic pain. development of physical factors.

It is stated that after arthroplasty surgery, besides the physiological factors, the factors related to the individuals may affect the recovery. Among these factors, one of the most defined in the literature is kinesiophobia. Although kinesiophobia is defined as the terms of "fear of movement" and "fear related to pain"; There are also definitions for situations in which fear of movement is most extreme or pain-related fear avoidance beliefs. Kinesiophobia, which usually occurs in the preoperative period and supports the development of chronic pain, may also affect the early recovery findings. It is very important to determine the presence and severity of kinesiophobia as it is associated with functional results after surgery.

Individuals' perceptions about themselves, expectations of recovery, and personal beliefs before surgery are thought to affect recovery in the early period. In the studies conducted, it was stated that individuals with high perception about himself and the surgical process recover faster and return to activities. However, it is emphasized that studies should be conducted on the effect of individuals' personal factors such as self-efficacy, self-perception and their perspective on health on the healing process.

Investigation of factors affecting functional capacity, balance and mobility in individuals who have undergone total knee surgery with these approaches; Taking into account the perceptual problems that exist in addition to orthopedic problems, all problems in education are addressed holistically. Our work based on this idea; It is planned to investigate the factors affecting functional capacity, balance and mobility in individuals who have undergone total knee arthroplasty surgery.

In our study, between February 2020 and March 2020, Fırat University Training and Research Hospital, an orthopedic specialist will be diagnosed with osteoarthritis and patients who will undergo total knee arthroplasty surgery will be evaluated. Factors affecting patients' functional capacity, balance and mobility will be investigated.

From the patient records, as demographic features; patients' age, gender, body weight, height, hand (dominant hemisphere), profession and educational status, history of the disease will be taken. To our orthopedic evaluation form; muscle strength, range of motion, gait analysis, kinesiophobia, pain state, contracture state, obesity state, condition of intracapsular structures, etc. Information about will be obtained.

With these data, it will be investigated whether there is a change in the functional capacity, balance and mobility of patients, and which factors its balance depends on.

Individuals will be obtained from the individuals before surgery, 1 month after surgery and 3 months after surgery: TAMPA Kinesiophobia Scale, Lequesne knee osteoarthritis severity index, WOMAC scale and gait analysis evaluation data.

Statistical analysis of the study will be made with "Statistical Package for Social Sciences" (SPSS) Version IBM Statistic 20. Demographic data will be given as mean ± SD. Students t test will be used in continuous variables analysis, and Chi Square Test will be used to compare percentages. Differences below P value <0.05 will be considered meaningful.

ELIGIBILITY:
* Inclusion Criteria:

  * Between 30-90 years old,
  * Primary unilateral total knee replacement will be applied due to knee osteoarthritis,
  * Patients volunteering to participate in the study
* Exclusion Criteria:

  * Who have neurological (hemiplegia, parkinson, multiplsclerosis etc.) disease that will affect functional performance and balance,
  * Does not have cognitive function to allow active participation,
  * Having a severe psychiatric condition,
  * Severe vision and hearing loss,
  * Any other treatment other than medication,
  * Who have contralateral knee osteoarthritis (pain with activity 4/10 or higher),
  * Using drugs that can cause loss of balance,
  * With more than 5 cm length difference in the lower extremities,
  * Having undergone lower limb trauma or surgery in the past 1 year,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with arthroplasty recommended for knee osteoarthritis
Sampling Method: Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-03-15 (Estimated); Study Completion 2020-05-15 (Estimated)

PRIMARY OUTCOMES:
The Tampa Scale of Kinesiophobia | 2 weeks
  Evaluation will be done before surgery .Individuals' kinesiophobia will be evaluated
The Tampa Scale of Kinesiophobia | 1 mounth
  Evaluation will be done before surgery at the 1st month.Individuals' kinesiophobia will be evaluated
The Tampa Scale of Kinesiophobia | 3 Mounth
  Evaluation will be done before surgery at the 3st month. Individuals' kinesiophobia will be evaluated

SECONDARY OUTCOMES:
The Western Ontario and McMaster Universities Arthritis Index (WOMAC) | 2 weeks
  Evaluation will be done before surgery, Pain, joint stiffness and function data will be evaluated.
The Western Ontario and McMaster Universities Arthritis Index (WOMAC) | 1 mounth
  Evaluation will be done before surgery, at the 1st months. Pain, joint stiffness and function data will be evaluated.
The Western Ontario and McMaster Universities Arthritis Index (WOMAC) | 3 mounth
  Evaluation will be done before surgery, at the 3rd months. Pain, joint stiffness and function data will be evaluated.
Spatio-temporal gait | 2 weeks
  Evaluation will be done before surgery. The data will be made with the Win-Track walking platform.
Spatio-temporal gait | 1 mounth
  Evaluation will be done before surgery, at the 1st. The data will be made with the Win-Track walking platform.
Spatio-temporal gait | 3 mounth
  Evaluation will be done before surgery, at the 3rd months. The data will be made with the Win-Track walking platform.
Lequesne Index | 2 weeks
  Evaluation will be done before surgery. It is a 10-item scale consisting of 3 sections: pain / discomfort, daily life activities and maximum walking distance.
Lequesne Index | 1 mounth
  Evaluation will be done before surgery, at the 1st. It is a 10-item scale consisting of 3 sections: pain / discomfort, daily life activities and maximum walking distance.
Lequesne Index | 3 mounth
  Evaluation will be done before surgery, at the 3rd months. It is a 10-item scale consisting of 3 sections: pain / discomfort, daily life activities and maximum walking distance.
Hormone level of iris | 2 weeks
  Evaluation will be done before surgery.Blood samples will be taken into gel biochemistry tubes, as appropriate for analysis from patients. The blood collected will be centrifuged for 10 minutes at 3000 rpm and the serum will be separated and the obtained serums will be placed in ependorphic tubes in small portions and stored at -80 ° C until analysis. The levels of iris will be studied in accordance with the kit user manual using commercial ELISA (enzyme-linked immunosorbent assay) kits.
Hormone level of iris | 1 Mounth
  Evaluation will be done before surgery, at the 1st. Blood samples will be taken into gel biochemistry tubes, as appropriate for analysis from patients. The blood collected will be centrifuged for 10 minutes at 3000 rpm and the serum will be separated and the obtained serums will be placed in ependorphic tubes in small portions and stored at -80 ° C until analysis. The levels of iris will be studied in accordance with the kit user manual using commercial ELISA (enzyme-linked immunosorbent assay) kits.
Hormone level of iris | 3 Mounth
  Evaluation will be done before surgery, at the 3rd months. Blood samples will be taken into gel biochemistry tubes, as appropriate for analysis from patients. The blood collected will be centrifuged for 10 minutes at 3000 rpm and the serum will be separated and the obtained serums will be placed in ependorphic tubes in small portions and stored at -80 ° C until analysis. The levels of iris will be studied in accordance with the kit user manual using commercial ELISA (enzyme-linked immunosorbent assay) kits.

CONTACTS AND LOCATIONS:
Locations (1):
- Fırat Univerity Hospital, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palazzo C, Nguyen C, Lefevre-Colau MM, Rannou F, Poiraudeau S. Risk factors and burden of osteoarthritis. Ann Phys Rehabil Med. 2016 Jun;59(3):134-138. doi: 10.1016/j.rehab.2016.01.006. Epub 2016 Feb 19. PMID 26904959
- [Background] Başkurt Z, Ercan S, Parpucu Tİ, Başkurt F, Ünal M. Diz Osteoartriti Olan Hastalarda Kinezyobant Uygulamasının Kısa Dönem Etkileri. Spor Hekimliği Dergisi. 2017;52(4):146-54.
- [Background] Arendt-Nielsen L, Nie H, Laursen MB, Laursen BS, Madeleine P, Simonsen OH, Graven-Nielsen T. Sensitization in patients with painful knee osteoarthritis. Pain. 2010 Jun;149(3):573-581. doi: 10.1016/j.pain.2010.04.003. Epub 2010 Apr 24. PMID 20418016
- [Background] Grayson CW, Decker RC. Total joint arthroplasty for persons with osteoarthritis. PM R. 2012 May;4(5 Suppl):S97-103. doi: 10.1016/j.pmrj.2012.02.018. PMID 22632709
- [Background] Ekşioğlu E, Gürçay E. Total diz artroplastisi sonrasi rehabilitasyon. İstanbul Tıp Fakültesi Dergisi. 2014;76(1):16-21.
- [Background] Alsancak S, Altinkaynak H, Güner S. Sosyal Güvenlik Kurumu verilerine göre Türkiye'de hastaya özel yapılarak uygulanan profitez ve ortezlerin sayısal çeşitlilik analizi. Fizyoterapi Rehabilitasyon
- [Background] Lotke PA. Primary Total Knee: Standard Principles and Technique In: Murphy RAHaD, editor. Knee Arthroplasty Lippincott Williams & Wilkins, a Wolters Kluwer business 2009.
- [Background] Mizner RL, Petterson SC, Snyder-Mackler L. Quadriceps strength and the time course of functional recovery after total knee arthroplasty. J Orthop Sports Phys Ther. 2005 Jul;35(7):424-36. doi: 10.2519/jospt.2005.35.7.424. PMID 16108583
- [Background] Demir H, Çalış M. Diz artroplastisi rehabilitasyonu. Erciyes Medical Journal. 2002;24(4):194-201.
- [Background] Aktuğ BB. Total diz artroplastili hastaların fonksiyonel düzeyleri ile memnuniyet düzeyleri arasındaki ilişkinin incelenmesi: DEÜ Sağlık Bilimleri Enstitüsü; 2009.
- [Background] Morrey BF, Adams RA, Ilstrup DM, Bryan RS. Complications and mortality associated with bilateral or unilateral total knee arthroplasty. J Bone Joint Surg Am. 1987 Apr;69(4):484-8. PMID 3571305
- [Background] Peersman G, Laskin R, Davis J, Peterson MG, Richart T. Prolonged operative time correlates with increased infection rate after total knee arthroplasty. HSS J. 2006 Feb;2(1):70-2. doi: 10.1007/s11420-005-0130-2. PMID 18751850
- [Background] Geiger M, editor The Influence Of Psychological Factors On Reducing Recovery Time From Total Knee Replacement Surgery. Symposium; 2015. 45
- [Background] Guney-Deniz H, Irem Kinikli G, Caglar O, Atilla B, Yuksel I. Does kinesiophobia affect the early functional outcomes following total knee arthroplasty? Physiother Theory Pract. 2017 Jun;33(6):448-453. doi: 10.1080/09593985.2017.1318988. Epub 2017 May 8. PMID 28481125
- [Background] Kocic M, Stankovic A, Lazovic M, Dimitrijevic L, Stankovic I, Spalevic M, Stojiljkovic P, Milenkovic M, Stojanovic Z, Nikolic D. Influence of fear of movement on total knee arthroplasty outcome. Ann Ital Chir. 2015 Mar-Apr;86(2):148-55. PMID 25952608
- [Background] Lundberg M. Kinesiophobia Various Aspects of Moving with Musculoskeletal Pain 2006.
- [Background] Hanusch BC, O'Connor DB, Ions P, Scott A, Gregg PJ. Effects of psychological distress and perceptions of illness on recovery from total knee replacement. Bone Joint J. 2014 Feb;96-B(2):210-6. doi: 10.1302/0301-620X.96B2.31136. PMID 24493186